CLINICAL TRIAL: NCT00572260
Title: A Pilot Study of Daptomycin for Antimicrobial Prophylaxis in Patients Undergoing Cardiac Valve Replacement and Coronary Artery Bypass Grafting (CABG) Who Are at Increased Risk for Infection Due to Methicillin-resistant Staphylococcus Aureus (MRSA)
Brief Title: A Pilot Study of Daptomycin for Antimicrobial Prophylaxis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study closed. PI left the institution.
Sponsor: Duke University (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Pro00000856; 19497
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2012-11

CONDITIONS: Antimicrobial Prophylaxis
Keywords: MRSA; Increased risk for infection
MeSH Terms: interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Daptomycin as a single preoperative dose within 30 minutes prior to surgery Dosage: if creatinine clearance ≥ 30 ml/min: 6 mg/kg IV
  Interventions: Drug: daptomycin 6 mg/kg IV

INTERVENTIONS:
Drug: daptomycin 6 mg/kg IV — daptomycin 6 mg/kg IV given during induction phase as a one-time prophylactic dose for patients undergoing cardiac valve replacement and coronary artery bypass grafting (CABG) who are at increased risk for infection due to methicillin-resistant Staphylococcus aureus (MRSA)

SUMMARY:
The goals of the study are to evaluate the feasibility of using daptomycin as a prophylactic antimicrobial agent in patients undergoing cardiac surgery, to determine the rates of surgical site infection, and to evaluate the occurrence of adverse events.

ELIGIBILITY:
INCLUSION CRITERIA: Patients will be eligible for inclusion in the study if they meet the following criteria:

1. Provide signed and dated informed consent and are willing to receive the study medication
2. Age ≥ 18 years of age
3. If a female of childbearing potential is willing to practice at least one method of birth control during treatment and for at least 28 days after treatment with study medication:

   1. barrier methods of birth control (e.g., condoms, diaphragms together with spermicidal foam or gel, or presence of IUD) or
   2. surgical sterilization, approved hormonal contraceptives (such as birth control pills, depo-Provera, or Lupron Depot), or IUD are all acceptable.

      * Rhythm, temperature, and verbal promise of abstinence are not acceptable methods of birth control.
4. If a female of childbearing potential, serum HCG negative within 24 hours of scheduled surgery.
5. Planned cardiac surgery procedures meeting current Duke criteria to receive anti-microbial prophylaxis active against MRSA:

   a. Patients will meet at least one of the following criteria which are the same as for prophylaxis with vancomycin: i. preoperative hospitalization > 48 hours ii. transfer to Duke from outside facility iii. previous history of MRSA iv. any patient deemed to be high risk for MRSA by the attending surgeon, due to a complicated past medical and/or surgical history

EXCLUSION CRITERIA: Patients who satisfy any of the following are not eligible for study enrollment.

1. Hypersensitivity to daptomycin
2. Inability to receive standard prophylaxis agents (cefuroxime and rifampin) for any reason
3. Staphylococcal bacteremia at the time of enrollment
4. Diagnosis of S. aureus or coagulase negative staphylococcus pacemaker/defibrillator infection within the preceding 18 months
5. Patient is undergoing emergency CABG
6. Weight >150 kg or <50kg
7. Patients considered unlikely to survive at least 7 days due to underlying illness.
8. Patients with creatinine clearance (CLcr) < 30mL/min (calculated using the Cockcroft-Gault equation using actual body weight)
9. Severe neutropenia (absolute neutrophil count <0.500x103 /µL)
10. Pregnant, nursing or lactating women (if patient is still of childbearing potential, a negative serum pregnancy test will be confirmed)
11. Patients considered unlikely to comply with study procedures or to return for the scheduled post treatment evaluation
12. Any other condition that in the opinion of an investigator, would confound or interfere with evaluation of safety or efficacy of the investigational medication, or prevent compliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith S Kaye, MD, MPH, Principal Investigator — DMC
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 1/17/2008 and 9/15/2008, 124 subjects were identified as qualifying, 56 were referred and approached, 44 refused to participate, and 12 signed the ICF at Duke University Hospital inpatient care units.
Pre-assignment Details: Between 1/17/2008 and 9/15/2008, among the 12 study subjects that signed the ICF, 11 subjects met the eligibility criteria and were enrolled in the study. One subject was disqualified due to weight > 150kg and was withdrawn from the study
Period: Overall Study
Arm/Group | Antimicrobial Prophylaxis Administration With Daptomycin
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Antimicrobial Prophylaxis Administration With Daptomycin
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Rate of Patients Receiving Antimicrobial Prophylaxis Within the Appropriate Timeframe Before Incision
Time Frame: 30 days after surgery
Population: The study closed due to the departure of the principal investigator and the data analysis was not performed.
Groups:
- Patients Undergoing Cardiac Surgery: Patients undergoing cardiac valve replacement and coronary artery bypass grafting
Arm/Group | Patients Undergoing Cardiac Surgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Antimicrobial Prophylaxis Administration With Daptomycin
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
Premature termination of the study due to departure of the PI resulted in falling short of enrollment goal (enrolled - 11 enrolled/goal - 100) leading to uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No